CLINICAL TRIAL: NCT06372210
Title: An Open-label, Prospective Trial Assessing Positive Detection Accuracy and Detection Latency Measures of the Miniature Ingestible Event Marker Tablet Using the D-Tect Patch in Healthy Subjects and Assessing Detection Latency Measures Using the D-Tect Patch in Subjects With Serious Mental Illness Taking Abilify MyCite Tablet
Brief Title: A Trial to Assess a Wearable Patch's Functioning to Detect Medication Ingestion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Otsuka Pharmaceutical Development & Commercialization, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 031-201-00521
Record Dates: First submitted 2024-03-29; First posted 2024-04-17 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Mental Disorder; Schizophrenia; Major Depressive Disorder; Bipolar I Disorder
Keywords: D-Tect patch
MeSH Terms: conditions — Mental Disorders; Schizophrenia; Depressive Disorder, Major

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- D-Tect Patch (Experimental): A D-Tect patch was applied by the clinical staff prior to each IEM tablet ingestion, and directly observed ingestions (DOIs), followed by ingestion of 15 placebo-embedded IEM tablets, 1 every 15 minutes in Cohort 1 on Day 1 and a single dose of Abilify MyCite® tablet in Cohort 2 on Day 1.
  Interventions: Drug: Placebo IEM tablet; Drug: Abilify MyCite®; Device: D-Tect Patch

INTERVENTIONS:
Drug: Placebo IEM tablet — Oral placebo-embedded IEM tablet.
Drug: Abilify MyCite® — Oral aripiprazole-embedded IEM tablet.
  Other Names: OPC-14597 Digital
Device: D-Tect Patch — The D-Tect patch is a wearable sensor (WS) capable of detecting the ingestion of the IEM and measuring physiologic parameters. The WS automatically logs and stores the time when the IEM reaches the stomach and transmits the data to a smartphone.

SUMMARY:
The primary purpose of the study is to evaluate the positive detection accuracy (PDA) and detection latency measures of the D-Tect patch.

DETAILED DESCRIPTION:
This is an open-label study to determine the accuracy of ingestible event marker (IEM) detection and detection latency of the D-Tect patch by completing a series of patch applications and IEM ingestions in the clinic.

The participants were enrolled in two cohorts within this study- Cohort 1: healthy participants received the placebo-embedded IEM tablets, Cohort 2: participants with serious mental illness (SMI) i.e schizophrenia, major depressive disorder, or bipolar I disorder received Abilify MyCite® tablets (aripiprazole-embedded IEM tablets).

This single-center trial was conducted in the United States. The overall time to participate in this study is up to approximately 17 days.

ELIGIBILITY:
Inclusion Criteria for Cohort 1:

* In good general health or medically stable.
* Is able and willing to participate in, and adhere to, all testing procedures, both onsite and offsite, for the entire testing.
* The participant has access to a telephone for communicating with the trial personnel and for trial personnel to contact the participant.

Inclusion Criteria for Cohort 2:

* In good general health or medically stable.
* Has confirmed diagnosis of schizophrenia, major depressive disorder, or bipolar I disorder per Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5) criteria and currently prescribed and taking aripiprazole.
* Is able and willing to participate in, and adhere to, all testing procedures, both onsite and offsite, for the entire testing.
* Participant has access to a telephone for communicating with the trial personnel and for trial personnel to contact the participant

Exclusion Criteria for Cohort 1 and 2:

* Any medical condition, treatment, or symptoms that, in the judgment of the trial clinician, could place the participant at more than the minimal risk from involvement in the testing.
* Hospitalization, emergency room visit, surgery or new medical treatment within 30 days before testing begins or planned during testing.
* Difficulty with or inability to swallow tablets.
* Active skin infection or active dermatitis, or history of chronic inflammatory skin condition including psoriasis and chronic dermatitis (except atopic dermatitis).
* The investigator will determine if any participant should be excluded from the trial based on history of, or current, alcohol abuse, drug abuse or use of illegal drugs (e.g., amphetamines or heroin).
* Allergy to adhesive bandages/tapes (e.g., Band-Aids®) or latex.
* Positive urine pregnancy test at screening visit (dipstick).
* Participant is taking any concomitant medication that places the participant at a greater risk for skin reactions or skin sensitivity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2023-06-26 (Actual); Primary Completion 2023-07-19 (Actual); Study Completion 2023-07-19 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Research site, Garden Grove, California, United States

IPD SHARING:
Plan to Share IPD: Yes
Anonymized Individual participant data (IPD) that underlie the results of this study will be shared with researchers to achieve aims pre-specified in a methodologically sound research proposal. Small studies with less than 25 participants are excluded from data sharing.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data will be available after marketing approval in global markets, or beginning 1-3 years following article publication. There is no end date to the availability of the data.
Access Criteria: Otsuka will share data on an Otsuka-owned remotely accessible data sharing platform with Python and R analytical software. Research requests should be directed to clinicaltransparency@Otsuka-us.com
URL: https://clinical-trials.otsuka.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at a single investigative site in the United States from 26 June 2023 to 19 July 2023.
Pre-assignment Details: A total of 54 participants were enrolled in this study and all participants completed the study.
Groups:
- Cohort 1: D-Tect Patch + Placebo-embedded IEM: A D-Tect patch was applied by the clinical staff prior to the first ingestion of a placebo-embedded ingestible event marker (IEM) tablet. Directly observed ingestions (DOIs) of 15 placebo-embedded IEM tablets were noted at 15-minute intervals on Day 1.
- Cohort 2: D-Tect Patch + Abilify MyCite® (Aripiprazole-embedded IEM): A D-Tect patch was applied by the clinical staff prior to the ingestion of the IEM-embedded Abilify MyCite® tablet. A DOI of a single dose of Abilify MyCite® tablet occurred on Day 1.
Period: Overall Study
Arm/Group | Cohort 1: D-Tect Patch + Placebo-embedded IEM | Cohort 2: D-Tect Patch + Abilify MyCite® (Aripiprazole-embedded IEM)
Started | 24 | 30
Completed | 24 | 30
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled analysis set included all participants who signed an informed consent form (ICF) and entered the study (and only participants who met all the inclusion criteria and none of the exclusion criteria).
Groups:
- Cohort 1: D-Tect Patch + Placebo-embedded IEM: A D-Tect patch was applied by the clinical staff prior to the first ingestion of a placebo-embedded IEM tablet. DOIs of 15 placebo-embedded IEM tablets were noted at 15 minute intervals on Day 1.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: D-Tect Patch + Placebo-embedded IEM | Cohort 2: D-Tect Patch + Abilify MyCite® (Aripiprazole-embedded IEM) | Total
Number analyzed (Participants) | 24 | 30 | 54
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.8 (13.56) | 46.1 (12.03) | 48.2 (12.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 10 | 27
  Male | 7 | 20 | 27
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 16 | 20
  Not Hispanic or Latino | 20 | 14 | 34
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 0
  Race: Asian | 12 | 1 | 13
  Race: Black or African American | 6 | 9 | 15
  Race: Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Race: White | 6 | 20 | 26
  Race: Other | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 24 | 30 | 54

OUTCOME MEASURES:

1. Primary Outcome: Cohort 1: Positive Detection Accuracy (PDA) of D-Tect Patch
Description: The PDA is calculated as the number of total positive detections by patch divided by the number of the total DOIs. PDA was estimated by Clopper-Pearson method.
Time Frame: At Day 1
Population: Full analysis set (FAS) comprised of all the detections of the wearable sensors done on the participants who took at least 1 dose of a miniature ingestible tablet (MIT) (Cohort 1), excluding those detections with device malfunction (invalid session and bad impedance). 'Overall number of participants analyzed' indicates the number of participants with at least one detection in Cohort 1.
Measure: Number (95% Confidence Interval); unit: percentage of detections
Units Other Than Participants: Number of detections
Arm/Group | Cohort 1: D-Tect Patch + Placebo-embedded IEM
Number analyzed (Participants) | 24
Number analyzed (Number of detections) | 358
percentage of detections | 100 [98.97 to 100]

2. Primary Outcome: Cohort 1 and 2: Patch Detection Latency Period
Description: The patch detection latency period is defined as the time between the ingestion of the tablet and the detection of the tablet ingestion by the patch. Kaplan Meier estimation was used to measure the patch detection latency period.
Time Frame: At Day 1
Population: The FAS comprised of all the detections of the wearable sensors done on the participants who took at least 1 dose of MIT (Cohort 1) or Abilify MyCite® (Cohort 2), excluding those detections with device malfunction (invalid session and bad impedance). "Overall number of participants analyzed" indicates the number of participants with at least one detection.
Measure: Median (Full Range); unit: seconds
Units Other Than Participants: Number of detections
Arm/Group | Cohort 1: D-Tect Patch + Placebo-embedded IEM | Cohort 2: D-Tect Patch + Abilify MyCite® (Aripiprazole-embedded IEM)
Number analyzed (Participants) | 24 | 30
Number analyzed (Number of detections) | 358 | 30
seconds | 53.0 [11 to 206] | 312.0 [90 to 695]

3. Primary Outcome: Cohort 1 and 2: Ingestion Data Transfer Latency Period
Description: The ingestion data transfer latency period is measured as the time between the detection of the tablet ingestion by the patch and the display of ingestion data on the mobile device. Kaplan Meier estimation was used to measure the ingestion data transfer latency period.
Time Frame: At Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: seconds
Units Other Than Participants: Number of detections
Arm/Group | Cohort 1: D-Tect Patch + Placebo-embedded IEM | Cohort 2: D-Tect Patch + Abilify MyCite® (Aripiprazole-embedded IEM)
Number analyzed (Participants) | 24 | 30
Number analyzed (Number of detections) | 358 | 30
seconds | 17.0 [0 to 536] | 17.0 [6 to 145]

4. Primary Outcome: Cohort 1 and 2: Total Detection Latency Period
Description: The total detection latency is measured as the total time between the ingestion of the tablet and the display of ingestion data on the mobile device. Kaplan Meier estimation was used to measure the total detection the latency period.
Time Frame: At Day 1
Population: as for outcome 2
Measure: Median (Full Range); unit: seconds
Units Other Than Participants: Number of detections
Arm/Group | Cohort 1: D-Tect Patch + Placebo-embedded IEM | Cohort 2: D-Tect Patch + Abilify MyCite® (Aripiprazole-embedded IEM)
Number analyzed (Participants) | 24 | 30
Number analyzed (Number of detections) | 358 | 30
seconds | 73.0 [11 to 587] | 351.0 [107 to 729]

5. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Device-related TEAEs, Serious TEAEs (SAEs), TEAEs Leading to Study Discontinuation
Description: TEAEs were defined as AEs that occurred on or after the participant wears any patch or takes any tablet from the study at test day, and the AEs that occurred before the participant wears any patch or takes any tablet and are worsening, serious, related, or resulted in death, discontinuation, or interruption of investigational product. A serious TEAE was defined as a TEAE that is fatal, life-threatening, results in persistent or significant disability/incapacity, constitutes a congenital anomaly/birth defect, or requires inpatient hospitalization or prolongation of existing hospitalization.
Time Frame: From Day 1 up to follow-up (up to Day 10)
Population: Safety analysis set included all participants who wore any patch or took any tablet from the study and had any safety assessment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: D-Tect Patch + Placebo-embedded IEM | Cohort 2: D-Tect Patch + Abilify MyCite® (Aripiprazole-embedded IEM)
Number analyzed (Participants) | 24 | 30
Participants
  Participants With TEAEs | 7 | 3
  Participants With Device-related TEAEs | 5 | 3
  Participants With Serious TEAEs | 0 | 0
  Participants With TEAEs Leading to Study Discontinuation | 0 | 0

ADVERSE EVENTS:
Time Frame: From Day 1 up to follow-up (up to Day 10)
Description: Safety analysis set included all participants who wore any patch or took any tablet from the study and had any safety assessment.
Arm/Group | Cohort 1: D-Tect Patch + Placebo-embedded IEM | Cohort 2: D-Tect Patch + Abilify MyCite® (Aripiprazole-embedded IEM)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/30
Other Adverse Events (participants affected / at risk) | 7/24 | 3/30
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: D-Tect Patch + Placebo-embedded IEM (N=24) | Cohort 2: D-Tect Patch + Abilify MyCite® (Aripiprazole-embedded IEM) (N=30)
Medical device site pruritus (General disorders) | 4 | 2
Medical device site erythema (General disorders) | 0 | 1
Medical device site irritation (General disorders) | 1 | 0
Faeces discoloured (Gastrointestinal disorders) | 0 | 1
Cheilitis (Gastrointestinal disorders) | 1 | 0
Nausea (Gastrointestinal disorders) | 1 | 0
Headache (Nervous system disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/10/NCT06372210/Prot_000.pdf
  • Statistical Analysis Plan (2023-06-22): https://cdn.clinicaltrials.gov/large-docs/10/NCT06372210/SAP_001.pdf